CLINICAL TRIAL: NCT04248855
Title: A Phase 1 Study of the Safety and Tolerability of Single and Multiple Doses of KAN-101 in Patients With Celiac Disease (ACeD)
Brief Title: Assessment of KAN-101 in Celiac Disease (ACeD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kanyos Bio, Inc., a wholly-owned subsidiary of Anokion SA (Industry)
Responsible Party: Sponsor
Organization: Anokion SA (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: KAN-101-01
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Celiac Disease
Keywords: Phase 1; Double blind; Multicenter
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- SAD Cohort 1 (Experimental): All enrolled patients will receive one dose of KAN-101 Dose A
  Interventions: Drug: KAN-101
- SAD Cohort 2 (Experimental): All enrolled patients will receive one dose of KAN-101 Dose B
  Interventions: Drug: KAN-101
- SAD Cohort 3 (Experimental): All enrolled patients will receive one dose of KAN-101 Dose C
  Interventions: Drug: KAN-101
- SAD Cohort 4 (Experimental): All enrolled patients will receive one dose of KAN-101 Dose D
  Interventions: Drug: KAN-101
- MAD Cohort 5 (Experimental): All randomized patients will receive 3 doses of either KAN-101 Dose A or placebo
  Interventions: Drug: KAN-101; Drug: Placebo
- MAD Cohort 6 (Experimental): All randomized patients will receive 3 doses of either KAN-101 Dose B or placebo
  Interventions: Drug: KAN-101; Drug: Placebo
- MAD Cohort 7 (Experimental): All randomized patients will receive 3 doses of either KAN-101 Dose C or placebo
  Interventions: Drug: KAN-101; Drug: Placebo

INTERVENTIONS:
Drug: KAN-101 — Intravenous (IV) infusion
Drug: Placebo — Intravenous (IV) infusion
  Arms: MAD Cohort 5; MAD Cohort 6; MAD Cohort 7

SUMMARY:
A safety study of KAN-101 in patients with celiac disease. The study has two parts:

1. Part A - first in human study in which patients receive a single dose of KAN-101
2. Part B - patients will receive three doses of either KAN-101 or placebo

DETAILED DESCRIPTION:
Study KAN-101-01 is a Phase 1, FIH study designed to evaluate the safety and tolerability of KAN-101 in patients with celiac disease on a gluten free diet (GFD).

An overview of the two parts and proposed dose groups is given below:

1. Part A (SAD): Patients will receive a single dose of KAN-101.
2. Part B (MAD): Patients will receive three doses of either KAN-101 or placebo.

ELIGIBILITY:
Key Inclusion Criteria:

1. Adults aged 18 to 70 years inclusive
2. Diagnosed with celiac disease based on positive serology (eg, tissue transglutaminase IgA antibody and/or deamidated gliadin peptide IgG) and intestinal histology consistent with ≥ Marsh Type II or with evidence of villous atrophy
3. Has HLA-DQ2.5 genotype (HLA-DQA1*05 and HLA-DQB1*02) (homozygotes or heterozygotes)
4. Has followed a GFD for > 12 months immediately prior to study entry
5. Negative or weak positive for tTG-IgA and negative or weak positive for DGP-IgA/IgG during screening
6. Male or female. Females of childbearing potential must use at least 2 acceptable birth control methods
7. Capable of understanding and complying with protocol requirements
8. Patient understands and has signed the informed consent form

Key Exclusion Criteria:

1. Refractory celiac disease
2. Selective IgA deficiency
3. Positive for HLA-DQ8 (DQA1*03, DQB1*0302)
4. Previous treatment with tolerance-inducing therapies for celiac disease
5. Known wheat allergy
6. Part B only: History of hyperacute or prolonged symptoms following gluten exposure
7. Uncontrolled or significant medical conditions (including active infections or chronic hepatitis) which, in the opinion of the Investigator, preclude participation
8. History of dermatitis herpetiformis
9. Pregnant or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Kanyos Bio, Inc.
Locations (13):
- United States (13):
  - Anaheim Clinical Trials, Anaheim, California
  - Diablo Clinical Research, Walnut Creek, California
  - Innovative Medical Research of South Florida, Aventura, Florida
  - GCP Research, St. Petersburg, Florida
  - Tandem Clinical Research, Marrero, Louisiana
  - Parexel International- EPCU Baltimore, Baltimore, Maryland
  - West Michigan Clinical Research Center, Wyoming, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Celiac Disease Center at Columbia University, New York, New York
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Aventiv Research, Columbus, Ohio
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Advanced Clinical Research, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murray JA, Wassaf D, Dunn K, Arora S, Winkle P, Stacey H, Cooper S, Goldstein KE, Manchanda R, Kontos S, Grebe KM. Safety and tolerability of KAN-101, a liver-targeted immune tolerance therapy, in patients with coeliac disease (ACeD): a phase 1 trial. Lancet Gastroenterol Hepatol. 2023 Aug;8(8):735-747. doi: 10.1016/S2468-1253(23)00107-3. Epub 2023 Jun 14. PMID 37329900

RESULTS

PARTICIPANT FLOW:
Groups:
- SAD 0.15mg/kg: All enrolled patients received one dose of 0.15mg/kg KAN-101
  KAN-101: Intravenous (IV) infusion
- SAD 0.3mg/kg: All enrolled patients received one dose of 0.3mg/kg KAN-101
  KAN-101: Intravenous (IV) infusion
- SAD 0.6mg/kg: All enrolled patients received one dose of 0.6mg/kg KAN-101
  KAN-101: Intravenous (IV) infusion
- SAD 1.2mg/kg: All enrolled patients received one dose of 1.2mg/kg KAN-101
  KAN-101: Intravenous (IV) infusion
- SAD 1.5mg/kg: All enrolled patients received one dose of 1.5mg/kg KAN-101
  KAN-101: Intravenous (IV) infusion
- MAD 0.15mg/kg: All randomized patients received 3 doses of 0.15mg/kg KAN-101
  KAN-101: Intravenous (IV) infusion
- MAD 0.3mg/kg: All randomized patients received 3 doses of 0.3mg/kg KAN-101
  KAN-101: Intravenous (IV) infusion
- MAD 0.6mg/kg: All randomized patients received 3 doses of 0.6mg/kg KAN-101
  KAN-101: Intravenous (IV) infusion
- MAD Placebo: All randomized patients received 3 doses of placebo
  Placebo: Intravenous (IV) infusion
Period: Overall Study
Arm/Group | SAD 0.15mg/kg | SAD 0.3mg/kg | SAD 0.6mg/kg | SAD 1.2mg/kg | SAD 1.5mg/kg | MAD 0.15mg/kg | MAD 0.3mg/kg | MAD 0.6mg/kg | MAD Placebo
Started | 4 | 3 | 3 | 3 | 1 | 6 | 7 | 8 | 6
Completed | 4 | 3 | 3 | 3 | 1 | 6 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- SAD 0.15mg/kg: All enrolled patients will receive one dose of 0.15mg/kg KAN-101
  KAN-101: Intravenous (IV) infusion
- SAD 0.3mg/kg: All enrolled patients will receive one dose of 0.3mg/kg KAN-101
  KAN-101: Intravenous (IV) infusion
- SAD 0.6mg/kg: All enrolled patients will receive one dose of 0.6mg/kg KAN-101
  KAN-101: Intravenous (IV) infusion
- SAD 1.2mg/kg: All enrolled patients will receive one dose of 1.2mg/kg KAN-101
  KAN-101: Intravenous (IV) infusion
- SAD 1.5mg/kg: All enrolled patients will receive one dose of 1.5mg/kg KAN-101
  KAN-101: Intravenous (IV) infusion
- MAD 0.15mg/kg: All randomized patients will receive 3 doses of 0.15mg/kg KAN-101
  KAN-101: Intravenous (IV) infusion
- MAD 0.3mg/kg: All randomized patients will receive 3 doses of 0.3mg/kg KAN-101
  KAN-101: Intravenous (IV) infusion
- MAD 0.6mg/kg: All randomized patients will receive 3 doses of 0.6mg/kg KAN-101
  KAN-101: Intravenous (IV) infusion
- MAD Placebo: All randomized patients will receive 3 doses of placebo
  Placebo: Intravenous (IV) infusion
- Total: Total of all reporting groups
Arm/Group | SAD 0.15mg/kg | SAD 0.3mg/kg | SAD 0.6mg/kg | SAD 1.2mg/kg | SAD 1.5mg/kg | MAD 0.15mg/kg | MAD 0.3mg/kg | MAD 0.6mg/kg | MAD Placebo | Total
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 1 | 6 | 7 | 8 | 6 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (19.05) | 30.3 (15.72) | 35.3 (9.29) | 29.3 (11.37) | 46 (0) | 47.2 (12.32) | 40.7 (10.69) | 36.3 (16.19) | 30.3 (10.88) | 38 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 1 | 1 | 5 | 5 | 7 | 3 | 31
  Male | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 1 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 3 | 3 | 3 | 1 | 6 | 7 | 8 | 6 | 41
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 3 | 3 | 1 | 6 | 7 | 8 | 6 | 41

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Treatment-emergent Adverse Events (TEAEs)
Description: Incidence and severity of treatment-emergent adverse events (TEAEs) as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 or higher
Time Frame: Up to 28 Days
Population: All patients who received any amount of study drug with treatment group based on the dose level received.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD 0.15mg/kg | SAD 0.3mg/kg | SAD 0.6mg/kg | SAD 1.2mg/kg | SAD 1.5mg/kg | MAD 0.15mg/kg | MAD 0.3mg/kg | MAD 0.6mg/kg | MAD Placebo
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 1 | 6 | 7 | 8 | 6
Participants
  TEAE | 4 | 3 | 2 | 3 | 1 | 6 | 5 | 7 | 4
  Grade 3 or higher TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  no TEAE | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2

2. Secondary Outcome: Cmax
Description: Geometric mean of maximum drug concentration (Cmax)
Time Frame: 0, 7, 15, 30, 60, 120, 180, 240, 300, 360 minutes post dose on Days 1 and and 7
Population: All patients who received at least 1 dose of KAN-101 and have at least 1 drug concentration value. A patient may have been excluded from summary statistics due to insufficient data or failure to meet acceptability criteria
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | SAD 0.15mg/kg | SAD 0.3mg/kg | SAD 0.6mg/kg | SAD 1.2mg/kg | SAD 1.5mg/kg | MAD 0.15mg/kg | MAD 0.3mg/kg | MAD 0.6mg/kg
Number analyzed (Participants) | 4 | 2 | 2 | 3 | 1 | 5 | 7 | 8
ng/mL
  Day 1 | 839 (498) | 1796 (1443) | 10900 (1140) | 19470 (3336) | 22350 | 967 (917) | 2527 (1299) | 5753 (1623)
  Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 6 | 7
  Day 7 |  |  |  |  |  | 588 (375) | 2937 (1539) | 6609 (754.7)

3. Secondary Outcome: AUC Last
Description: Area under the plasma concentration-time curve from time 0 to the last measurable time point (AUC last)
Time Frame: 0, 7, 15, 30, 60, 120, 180, 240, 300, 360 minutes post dose on Days 1 and and 7
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SAD 0.15mg/kg | SAD 0.3mg/kg | SAD 0.6mg/kg | SAD 1.2mg/kg | SAD 1.5mg/kg | MAD 0.15mg/kg | MAD 0.3mg/kg | MAD 0.6mg/kg
Number analyzed (Participants) | 3 | 2 | 2 | 3 | 1 | 5 | 7 | 8
h*ng/mL
  Day 1 | 366.8 (147.7) | 646.3 (526.7) | 5365 (62.85) | 13920 (3033) | 16340 | 322.5 (290.7) | 1180 (653.7) | 3462 (986.4)
  Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 6 | 7
  Day 7 |  |  |  |  |  | 205 (152) | 1258 (751) | 3914 (760)

ADVERSE EVENTS:
Time Frame: Up to 28 Days
Arm/Group | SAD 0.15mg/kg | SAD 0.3mg/kg | SAD 0.6mg/kg | SAD 1.2mg/kg | SAD 1.5mg/kg | MAD 0.15mg/kg | MAD 0.3mg/kg | MAD 0.6mg/kg | MAD Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 0/3 | 0/1 | 0/6 | 0/7 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 0/3 | 0/1 | 0/6 | 0/7 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 2/3 | 3/3 | 1/1 | 6/6 | 5/7 | 7/8 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAD 0.15mg/kg (N=4) | SAD 0.3mg/kg (N=3) | SAD 0.6mg/kg (N=3) | SAD 1.2mg/kg (N=3) | SAD 1.5mg/kg (N=1) | MAD 0.15mg/kg (N=6) | MAD 0.3mg/kg (N=7) | MAD 0.6mg/kg (N=8) | MAD Placebo (N=6)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 4 (13) | 1 (3) | 3 (4) | 1 (5) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (7) | 2 (3) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 2 (3) | 2 (3) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 3 (3) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (6) | 1 (2) | 2 (2) | 1 (1) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 1 (1) | 1 (3) | 1 (1) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 1 (1) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Feeling Cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Cold Sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Abdominal Tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Aphthous Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Frequent Bowel Movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Steatorrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Feeling Hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Peripheral Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal
Eye Pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Treatment-Emergent Adverse Events Related to Investigational Medicinal

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/55/NCT04248855/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT04248855/SAP_001.pdf